CLINICAL TRIAL: NCT05378594
Title: Nasal Allergen Challenge: Standardisation for House Dust Mite and Silver Birch Allergen Extracts
Brief Title: HDM and Silver Birch NAC Standardisation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Royal Brompton & Harefield NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 84388
Record Dates: First submitted 2022-05-12; First posted 2022-05-18 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Intervention Model Description: 20 participants with silver birch pollen allergic rhinitis, 20 with house dust mite allergic rhinitis, dual allergic participants will be able to take part in both arms of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- House dust mite nasal allergen challenge (Experimental): House dust mite allergic patients to undergo nasal allergen challenge with house dust mite extract
  Interventions: Diagnostic Test: Nasal allergen challenge
- Silver birch pollen nasal allergen challenge (Experimental): Silver birch pollen allergic patients to undergo nasal allergen challenge with silver birch pollen extract
  Interventions: Diagnostic Test: Nasal allergen challenge

INTERVENTIONS:
Diagnostic Test: Nasal allergen challenge — graded nasal allergen challenge to increasing concentrations of allergen with monitoring of nasal symptoms and peak nasal inspiratory flow

SUMMARY:
This study aims to establish dose-responses to nasal allergen challenge using silver birch pollen and house dust mite allergen extracts in participants with allergic rhinitis, sensitised to either or both of these allergens. The allergen extracts used will be Itulazax tablets (silver birch pollen allergen sublingual tablets, ALK-Abello, Denmark) and Acarizax tablets (house dust mite allergen sublingual tablets, ALK-Abello, Denmark). The results will allow identification of the dose of each allergen typically producing a moderate severity response, which could then be used in future, interventional and investigational studies.

A control group - healthy individuals with no allergic rhinitis - will be recruited to demonstrate the absence of an irritant/non-allergic effect of the nasal allergen challenge procedure.

DETAILED DESCRIPTION:
Nasal allergen challenge (NAC) is a useful tool in the investigation of allergic rhinitis, including grass pollen-induced seasonal allergic rhinitis (hay fever). The investigators have experience in using NAC to investigate the clinical and immunological effects of allergen exposure and in using NAC as a surrogate outcome to assess the efficacy of treatments for allergic rhinitis. The procedure is safe and well tolerated.

For NAC to be a valid tool, it is essential that the allergen extracts used are standardised in terms of concentration and stability in solution. The investigators recently undertook a study comparing the effects of two different grass pollen allergen extracts when used for NAC. The investigators found that the use of a lyophilizate pollen tablet, designed for sublingual immunotherapy treatment, was a suitable alternative to using dissolved dry powder allergen, designed for subcutaneous immunotherapy treatment. The study was necessary because the dry powder product was being phased out by the manufacturer.

The investigators now intend to undertake a similar study using lyophilizate tablets for two further common environmental allergens, house dust mite and silver birch tree pollen. The products used will be as follows: Acarizax® House Dust Mite lyophilizate tablet and Itulazax® Silver Birch Pollen lyophilizate tablet, both manufactured by ALK-Abello, Denmark.

House dust mite (HDM) is the most common indoor allergen trigger in individuals with allergic rhinitis and allergic asthma in the UK; silver birch (SB) pollen is a common cause of springtime hay fever. This will allow us to determine the suitability of using lyophilizate tablets as an allergen source for NAC for these two allergens in future interventional studies.

In this study, the investigators will recruit 20 volunteers with house dust mite induced allergic rhinitis (+/- controlled asthma) and 20 volunteers with silver birch pollen induced allergic rhinitis (+/- controlled asthma); individuals allergic to both allergens will be eligible for both parts of the study. HDM allergic volunteers will undergo a graded, up-dosing NAC with HDM allergen tablet extract; SB allergic volunteers will undergo a graded, up-dosing NAC with SB allergen tablet extract; dual allergic individuals will be given the option of undergoing challenges to both allergens, at least 4 weeks apart.

Recorded outcomes will include the participant-reported symptom score (total nasal symptom score, TNSS, range 0-12) and peak nasal inspiratory flow (PNIF, L/min) during the NAC. The primary endpoint will be the area under the curve for TNSS during NAC with each allergen. Secondary endpoints will include area under the curve for change from baseline PNIF during NAC, the modal allergen dose required to give a TNSS of 7/12 ('provoking dose 7' ), peak TNSS score, maximal % fall in PNIF, and the absolute sneeze count.

Following the above, the investigators will then undertake nasal challenges using the identified 'provoking dose 7' for each allergen on 5 individuals from the other part of the cohort (i.e. test the HDM 'provoking dose 7' on 5 of the participants with SB allergy but no HDM allergy and vice versa) and also on 5 non-atopic individuals (no history of allergic rhinitis or asthma, negative skin tests to common environmental allergens), to prove the NAC is allergen specific and non-irritant.

The study will have two arms, one for HDM allergic individuals, one for SB allergic individuals, running concurrently. Dual allergic individuals may be included in both arms. Within each arm, up to 20 participants will undergo NAC with the relevant allergen. The NAC procedure will involve baseline TNSS and PNIF scores prior to intervention, then the same scores at 10 minutes after challenges with allergen at the following concentrations: 0 BU/mL (saline 1); 0 BU/mL (saline 2); 100 BU/mL; 500 BU/mL; 1,500 BU/mL; 5,000 BU/mL; 10,000 BU/mL, with 15 minutes between doses. Area under the curve for TNSS will be calculated for each NAC, along with the first concentration provoking a TNSS of ≥7/12. The NAC will continue to the top concentration of 10,000 BU/mL regardless of TNSS score, unless the participant has very bothersome symptoms and prefers not to continue.

For individuals allergic to both allergens, a minimum gap of 4 weeks will be required between the two NACs.

Following completion of the above and identification of the 'provoking dose 7' for each allergen, 5 single-sensitised (i.e. HDM or SB but not both) participants will return for a further NAC with the allergen to which they are not sensitised (a minimum of 4 weeks after their last NAC). The procedure will involve baseline TNSS and PNIF scores prior to intervention, then the same scores at 10 minutes after challenges with allergen at the following concentrations: 0 BU/mL (saline 1); 'provoking dose 7' BU/mL. Additionally, 5 non-atopic individuals will be recruited to attend for a single visit for NAC as follows: 0 BU/mL (saline 1); 'provoking dose 7' for HDM BU/mL; 0 BU/mL (saline 2); 'provoking dose 7' for SB BU/mL, with TNSS and PNIF measured as before.

Individuals with a history of seasonal allergic rhinitis in February-May and/or a history of perennial allergic rhinitis, suspected to be provoked by house dust mite exposure, for at least the past two years, will be invited for screening. Volunteers will need to avoid taking antihistamines for 5 days prior to screening to allow for skin testing. Up to forty volunteers (fewer if individuals are dual allergic and wish to take part in both arms of the study) who pass the inclusion and exclusion criteria (see below) and are willing to provide written, informed consent will be enrolled into the study. A minimum of five non-atopic individuals with no history of rhinitis who pass the inclusion and exclusion criteria (see below) will be enrolled into the control arm of the study. They will then undertake a single visit, as above.

Single allergen allergic individuals will undertake 1-2 visits after screening: Visit 1, all, challenge to relevant allergen; Visit 2, a minimum of 5, challenge to irrelevant allergen.

Dual allergen allergic individuals will undertake 1-2 visits after screening: Visit 1, all, challenge to allergen identified by participant and study doctor as the primary cause of their symptoms; Visit 2, as per participants preference, challenge to the other allergen.

Non-atopic volunteers will undertake a single visit after screening.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria (HDM allergic volunteers):

  1. Adults aged 18 to 65 years
  2. A clinical history of perennial allergic rhinitis for at least 2 years with house dust mite allergen a potential cause of symptoms
  3. Positive skin prick test response, defined as wheal diameter ≥ 5 mm, to house dust mite allergen extract
  4. For women of childbearing age, a negative urine pregnancy test at the time of screening and willingness to use an effective form of contraception for the duration of involvement in the study.
  5. The ability to give informed consent and comply with study procedures.

Inclusion criteria (SB allergic volunteers):

1. Adults aged 18 to 65 years.
2. A clinical history of seasonal allergic rhinitis in February-May for at least 2 years.
3. Positive skin prick test response, defined as wheal diameter ≥ 5 mm, to silver birch pollen allergen extract.
4. For women of childbearing age, a negative urine pregnancy test at the time of screening and willingness to use an effective form of contraception for the duration of involvement in the study.
5. The ability to give informed consent and comply with study procedures.

Inclusion criteria for non-atopic controls

1. Adults aged 18 to 65 years.
2. The ability to give informed consent and comply with study procedures.

Exclusion Criteria:

* Exclusion criteria (allergic volunteers):

  1. History of previous allergen immunotherapy to the relevant allergen being tested in the past 10 years
  2. Pre-bronchodilator FEV1 < 70% of predicted value at screening.
  3. Perennial asthma requiring regular inhaled corticosteroids.
  4. History of emergency visit or hospital admission for asthma in the previous 12 months.
  5. History of chronic obstructive pulmonary disease
  6. History of significant recurrent acute sinusitis, defined as 2 episodes per year for the last 2 years, all of which required antibiotic treatment.
  7. History of chronic sinusitis, defined as sinus symptoms lasting greater than 12 weeks that includes 2 or more major factors or 1 major factor and 2 minor factors. Major factors are defined as facial pain or pressure, nasal obstruction or blockage, nasal discharge or purulence or discolored postnasal discharge, purulence in nasal cavity, or impaired or loss of smell. Minor factors are defined as headache, fever, halitosis, fatigue, dental pain, cough, ear pain, pressure, or fullness.
  8. At screening visit, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media, or other relevant infectious process; serous otitis media is not an exclusion criterion. Participants may be re-evaluated for eligibility after symptoms resolve.
  9. History of life-threatening anaphylaxis or angioedema.
  10. Ongoing systemic immunosuppressive treatment.
  11. The use of any investigational drug within 30 days of the screening visit.
  12. The presence of any medical condition that the investigator deems incompatible with participation in the study.

Exclusion criteria for non-atopic controls

1. A history of hay fever, chronic rhinitis/rhinosinusitis other than symptoms experienced during viral colds or other respiratory tract infections.
2. A positive skin prick test to any of a panel of common aeroallergens including grass pollen (Timothy grass), silver birch (Betula verrucosa), house dust mite (Dermatophagoides pteronyssinus), cat hair (Felis domesticus), dog hair (Canis familiaris), and common moulds (Aspergillus fumigatus., Cladosporium sp., Alternaria sp.), with adequate positive and negative controls.
3. Pre-bronchodilator FEV1 < 70% of predicted value at screening.
4. Perennial asthma requiring regular inhaled corticosteroids.
5. History of emergency visit or hospital admission for asthma in the previous 12 months.
6. History of chronic obstructive pulmonary disease
7. At screening visit, current symptoms of, or treatment for, upper respiratory tract infection, acute sinusitis, acute otitis media, or other relevant infectious process; serous otitis media is not an exclusion criterion. Participants may be re-evaluated for eligibility after symptoms resolve.
8. History of life-threatening anaphylaxis or angioedema.
9. Ongoing systemic immunosuppressive treatment.
10. The use of any investigational drug within 30 days of the screening visit.
11. The presence of any medical condition that the investigator deems incompatible with participation in the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2022-09-22 (Actual); Primary Completion 2022-12 (Estimated); Study Completion 2022-12 (Estimated)

PRIMARY OUTCOMES:
Total nasal symptom score, area under the curve, during nasal allergen challenge | 0-90 minutes
  0-12 scale

SECONDARY OUTCOMES:
Peak nasal inspiratory flow, area under the curve, during nasal allergen challenge | 0-90 minutes
  L/min

OTHER OUTCOMES:
Modal dose of allergen provoking a total nasal symptom score of at least 7/12 for each allergen | 10 minutes
  As above

CONTACTS AND LOCATIONS:
Overall Officials: Guy Scadding, MD PhD, Principal Investigator — Royal Bromtpton Hospital
Locations (1):
- Royal Brompton Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No